CLINICAL TRIAL: NCT06333626
Title: Effects of an Oral Multi-vitamin Carbohydrate Beverage on Intraoperative Nausea and Vomiting in Women Converted From Vaginal Delivery to Cesarean Section
Brief Title: Effects of an Oral Multi-vitamin Carbohydrate Beverage on Intraoperative Nausea and Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020281
Record Dates: First submitted 2024-03-13; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-12

CONDITIONS: Nausea and Vomiting, Aspiration, Intraoperative
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation group (Experimental)
  Interventions: Dietary Supplement: multi-vitamin carbohydrate
- Control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: multi-vitamin carbohydrate — oral multi-vitamin carbohydrate beverage
  Arms: Observation group

SUMMARY:
Nausea and vomiting are common and unpleasant symptoms for pregnant women during cesarean section, which can lead to aspiration, a serious complication that can cause pneumonia. Our study aimed to evaluate the effects of oral multi-vitamin carbohydrate beverage on maternal intraoperative nausea and vomiting by gastric ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* at least 37 weeks pregnant, had not eaten for at least 4 h before entering the delivery room, converted from vaginal delivery to cesarean section

Exclusion Criteria:

* gestational diabetes mellitus or gastroesophageal reflux disease, cesarean section performed under general anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Gastric antrum area | one hour after eating, two hours after eating, and before entering operating room
  The gastric antrum area measured by gastric ultrasound

SECONDARY OUTCOMES:
vomiting | During the cesarean section
  The number of times pregnant woman vomits during cesarean section
The pH of vomiting fluid | During the cesarean section
  The pH of vomiting fluid recorded by a pen pH meter